CLINICAL TRIAL: NCT00442806
Title: A Randomized Clinical Trial of AdiPOse-derived Stem ceLLs in the Treatment of Patients With ST-elevation myOcardial Infarction - The APOLLO Trial
Brief Title: Randomized Clinical Trial of Adipose-Derived Stem Cells in the Treatment of Pts With ST-elevation Myocardial Infarction
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cytori Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: APOLLO - 01
Record Dates: First submitted 2007-02-28; First posted 2007-03-02 (Estimated); Last update posted 2013-11-26 (Estimated); Status verified 2013-11

CONDITIONS: Myocardial Infarction; Coronary Arteriosclerosis; Cardiovascular Disease; Coronary Disease
Keywords: ADRC; Stem Cells; Myocardial Infarction; STEMI; Heart Disease; Coronary Artery Disease; Coronary Disease; ST-Elevation; AMI; Interventional Cardiology; Heart Attack
MeSH Terms: conditions — Myocardial Infarction; Coronary Artery Disease; Cardiovascular Diseases; Coronary Disease; ST Elevation Myocardial Infarction; Heart Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Placebo is injected
  Interventions: Other: Injection of Placebo
- Treatment (Experimental): ADRC's are injected
  Interventions: Drug: Injection of ADRC's

INTERVENTIONS:
Drug: Injection of ADRC's — ADRC's are injected
  Arms: Treatment
Other: Injection of Placebo — Placebo is injected
  Arms: Placebo

SUMMARY:
The purpose of this study is to establish safety and feasibility of utilizing Adipose-Derived Stem and Regenerative Cells (ADRC's) in patients who have suffered a ST-elevation acute myocardial infarction.

DETAILED DESCRIPTION:
Subjects who have coronary artery disease and have suffered a ST-elevation acute myocardial infarction will be evaluated for eligibility in this study. Eligible subjects will undergo standard treatment after admission to the hospital and will then undergo liposuction under local anesthesia, after which ADRC's will be isolated from the lipoaspirate. According to randomization subjects will receive either ADRC's or placebo.

ELIGIBILITY:
Key Inclusion Criteria:

* Acute myocardial infarction (AMI)
* Clinical symptoms consistent with AMI for a minimum of 2 and a maximum of 12 hours from onset of symptoms to Percutaneous Coronary Intervention (PCI), and unresponsive to nitroglycerin
* Successful revascularization of the culprit lesion in the major epicardial vessel
* Area of hypo- or akinesia corresponding to the culprit lesion, as determined by left ventriculogram at the time of primary PCI
* Left ventricular ejection fraction (LVEF) ≥30% and ≤50% by Left Ventricular Angiography at the time of successful revascularization.
* Ability to undergo liposuction

Key Exclusion Criteria:

* Prior MI, prior known cardiomyopathy, or prior hospital admission for congestive heart failure (CHF)
* More than 24 hours after acute PCI
* Significant valvular disease
* More than twelve hours between the onset of first symptoms of AMI and revascularization
* Hemodynamic instability within 24 hours prior to randomization
* Neoplasia
* Acute or chronic bacterial or viral infectious disease
* Pacemaker, ICD or any other contra-indication for MRI
* LVEF <30% or >50% by Left Ventricular Angiography
* Moderate or severe COPD

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2007-11; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Safety - Determined by Major Adverse Cardiac and Cerebral Events (MACCE) | 6 months

SECONDARY OUTCOMES:
Feasibility - Assessment of cardiac function via functional and imaging studies including MRI, SPECT, and Echocardiography | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Eric Duckers, MD, PhD, Principal Investigator — Erasmus University Medical Centrum, ThoraxCenter
Locations (2):
- Erasmus University Medical Centrum, Thorax Center, Rotterdam, Netherlands
- Hospital General Universitario Gregorio Maranon, Madrid, Spain